CLINICAL TRIAL: NCT06231212
Title: Efficacy of a Standardized Centella Asiatica Extract in Patients With Temporomandibular Disorder
Acronym: TMD ECa233
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Prangtip Potewiratnanond D.D.S, M.Sc., Ph.D., Dr., Chulalongkorn University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CRP6305031970
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Temporomandibular Disorder
Keywords: TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — ECa 233 extract; Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal; Lactose

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo- and active-controlled clinical trial was performed on 18 to 50-year-old participants with acute TMD. These were randomly assigned to four treatment groups for 14 days: placebo, ibuprofen, ECa 233 250mg and 500 mg. At baseline, subjects reported 5 to 8 (out of 10) of pain intensity on a numerical rating scale (NRS). No medications were self-reported 24 hours before and during the trial and no systemic conditions were diagnosed. Degenerative joint disease was screened before treatment. Pain intensity levels, mandibular range of motion including pain-free, unassisted and assisted mouth opening, were recorded at baseline and 7 and 14 days post-treatment. Masticatory muscle and jaw joint tenderness were evaluated upon palpation according to the Diagnostic Criteria for TMD (DC/TMD).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ECa groups (Experimental): Intervention group takes capsules containing of ECa 233, an active substance composed of Madecassoside and Asiaticoside
  Interventions: Drug: ECa 233
- NSAID group (Active Comparator): Active-controlled group was given capsules containing 200 mg of ibuprofen
  Interventions: Drug: Ibuprofen
- Placebo group (Placebo Comparator): Placebo-controlled group received capsules containing 250 mg of lactose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ECa 233 — Intervention groups are separated into group A and group B. Group A takes capsules containing 250 mg of ECa 233 and group B takes capsules containing 500 mg of ECa 233.
  Arms: ECa groups
Drug: Ibuprofen — Ibuprofen group was given capsules containing 200 mg of ibuprofen
  Other Names: NSAIDs
  Arms: NSAID group
Other: Placebo — Placebo-controlled group received capsules containing 250 mg of lactose
  Other Names: lactose
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to test analgesic effect of ECa 233 in subjects with TMD. The main questions it aims to answer are:

* Can ECa 233 reduce pain intensity score in subjects with acute TMD?
* Can ECa 233 increase jaw functional movements in subjects with acute TMD? Participants will be separated into four groups, including placebo, ibuprofen, low-dosed Eca and high-dosed Eca groups.

DETAILED DESCRIPTION:
ECa 233 is a standardized extract of Centella asiatica with known anti-inflammatory properties and an acceptable safety profile. Hence, it would be relevant to evaluate the anti-inflammatory and pain reducing effects of ECa 233 on subjects with acute TMD, as well as jaw functional movements. A randomized, double-blind, placebo- and active-controlled clinical trial was performed on 18 to 50-year-old participants with acute TMD. These were randomly assigned to four treatment groups for 14 days: placebo, ibuprofen, ECa 233 250mg and 500 mg. At baseline, subjects reported 5 to 8 of pain intensity on a numerical rating scale (NRS). No medications were self-reported 24 h before and during the trial and no systemic conditions were diagnosed. Degenerative joint disease was screened before treatment. Pain intensity levels, mandibular range of motion including pain-free, unassisted and assisted mouth opening at baseline and days7 and 14 post-treatment. Masticatory muscle and jaw joint tenderness were evaluated upon palpation.

ELIGIBILITY:
Inclusion criteria

* Subjects reporting TMD pain lasting for 30 days or less (acute pain)
* Subjects with pain ratings between 5 and 8 on a 0-10 numerical rating scale

Exclusion criteria

* Subjects with any underlying chronic disease
* Subjects undergo any sort of treatment that may influence pain perception and/or inflammation, including as diabetes, psychological distress, systemic inflammatory disorders, oral appliances, and medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of ECa 233 for pain intensity | 14 days
  The pain intensity self-reported levels and other clinical parameters were collected at 3 time points: pre-intervention (baseline), 7 and 14 days post-intervention. The pain intensity score was determined by using a 10-point ordinal scale (0 representing no pain and 10 indicating severe pain).
Efficacy of ECa 233 capsules for jaw function | 14 days
  Mandibular range of motion, including pain-free, unassisted and assisted mouth opening,
Clinical efficacy of ECa 233 capsules in reducing areas of pain on palpation | 14 days
  The number of masticatory muscles and TMJs with pain upon palpation were counted on the left and right sides. The total score ranged from 0-12 locations

CONTACTS AND LOCATIONS:
Overall Officials: Prangtip Potewiratnanond, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Derived] Potewiratnanond P, Surarit R, Tantisira MH, Samaranayake L, Rotpenpian N, Wanasuntronwong A. Efficacy of Centella asiatica on mitigating temporomandibular pain and improving functionality: a randomized, double blind, pilot clinical trial. Head Face Med. 2025 Apr 19;21(1):28. doi: 10.1186/s13005-025-00503-y. PMID 40253389